CLINICAL TRIAL: NCT03642951
Title: Multi-site Transcranial Magnetic Stimulation Therapy of the Supplementary Motor Area in Children With Tourette Syndrome
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Low Enrollment
Sponsor: Children's Mercy Hospital Kansas City (Other)
Collaborators: The Methodist Hospital Research Institute (Other); Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14050210
Record Dates: First submitted 2018-03-21; First posted 2018-08-22 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-01

CONDITIONS: Tourette Syndrome
Keywords: magnetic; brain; stimulation
MeSH Terms: conditions — Tourette Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Treatment Group (Active Comparator): Each patient will receive daily 40 min treatment five days per week for two weeks. The procedure during each treatment session will consist of positioning the device centered at 15% of the nasion-inion distance anterior to the Cz electrode placement in standard EEGs, with the patient relaxing in a chair.
  The stimulus parameters used will be 480 stimulus trains of 100 ms in duration, each train delivered every 5 s for total session duration of 40 min. The investigator will measure the subject for accurate placement of the device prior to each visit. Once the placement of the device is confirmed, the study technician administering the treatment will tum on the device using an app downloaded to an electronic device connected by Bluetooth to the device.
  Interventions: Device: Active Treatment
- Sham Treatment Group (Sham Comparator): Each patient will receive daily 40 min treatment five days per week for two weeks. The procedure during each treatment session will consist of positioning the device centered at 15% of the nasion-inion distance anterior to the Cz electrode placement in standard EEGs, with the patient relaxing in a chair.
  The stimulus parameters used will be 480 stimulus trains of 100 ms in duration, each train delivered every 5 s for total session duration of 40 min. The investigator will measure the subject for accurate placement of the device prior to each visit. Once the placement of the device is confirmed, the study technician administering the treatment will tum on the device using an app downloaded to an electronic device connected by Bluetooth to the device.
  Note: While the device looks and is operated the same as the active device, subjects in this group will be stimulated with the placebo device so no active stimulation will be given.
  Interventions: Device: Sham Treatment

INTERVENTIONS:
Device: Active Treatment — The study patients will be randomly assigned to two groups, each consisting of 10 patients: Group A - patients stimulated by devices marked A; Group B - patients stimulated by devices marked B. Since the devices used for actual and sham stimulation (placebo control) are similar in all respects including external appearance and the sound produced while activated, the technician(s), investigators and the patients will be completely blind to whether actual or sham stimuli are being delivered, i.e. whether Group A or Group B patients are receiving the actual stimuli. Indeed, both devices marked A&B could be used to deliver either type of stimuli. Only the person who constructed the devices will know which is which. Therefore, this study will be a truly randomized double-blinded placebo-controlled clinical trial. In case of emergency, un-blinding of the device will be available to the study team via a sealed envelope, stored with the study documents, separate from the subjects study files.
  Other Names: Transcranial Rotating Permanent Magnet Stimulator (TRPMS)
  Arms: Active Treatment Group
Device: Sham Treatment — The study patients will be randomly assigned to two groups, each consisting of 10 patients: Group A - patients stimulated by devices marked A; Group B - patients stimulated by devices marked B. Since the devices used for actual and sham stimulation (placebo control) are similar in all respects including external appearance and the sound produced while activated, the technician(s), investigators and the patients will be completely blind to whether actual or sham stimuli are being delivered, i.e. whether Group A or Group B patients are receiving the actual stimuli. Indeed, both devices marked A&B could be used to deliver either type of stimuli. Only the person who constructed the devices will know which is which. Therefore, this study will be a truly randomized double-blinded placebo-controlled clinical trial. In case of emergency, un-blinding of the device will be available to the study team via a sealed envelope, stored with the study documents, separate from the subjects study files.
  Other Names: Transcranial Rotating Permanent Magnet Stimulator (TRPMS) (SHAM)
  Arms: Sham Treatment Group

SUMMARY:
The investigators are investigating the effectiveness of a wearable multisite transcranial magnetic stimulation (mTMS) device that can deliver stimuli at multiple cortical sites simultaneously or sequentially for the treatment of Tourette Syndrome.

DETAILED DESCRIPTION:
STUDY OBJECTIVES/HYPOTHESIS

Tourette Syndrome (TS) is a neurodevelopmental condition that affects nearly 1% of children world-wide. While it can be treated with drugs and behavioral therapy, other modalities are being sought, especially, in cases that are resistant to standard treatment. One such approach that is being tested in pilot clinical studies is repetitive transcranial magnetic stimulation (rTMS). Noninvasive magnetic stimulation of the cerebral cortex is an important and useful technique in neuroscience research, as well as in diagnostic and therapeutic clinical investigations. Over the last three decades the magnetic stimulation procedure is being carried out using a device called transcranial magnetic stimulator (TMS), which uses a large hand-held electromagnetic coil passing high amplitude current to induce a rapidly changing magnetic field at a single cortical site. TMS has found clinical application in several neurological and psychiatric conditions such as stroke, major depression, migraine, movement disorders and Tourette syndrome. One limitation of conventional TMS, besides the bulkiness of the device and the large amount of current involved, is that it allows stimulation at only one cortical site at a time. Dr. Santosh Helekar of Houston Methodist Research Institute (HMRI) and Dr. Henning Voss of Weill-Cornell Medical College (WCMC) have developed a compact portable and wearable multisite transcranial magnetic stimulation (mTMS) device that can deliver stimuli at multiple cortical sites simultaneously or sequentially. It uses rapidly rotating small high strength permanent magnets to induce currents in the brain. As opposed to conventional TMS, the mTMS device is also ideally suited to conduct double-blind placebo-controlled studies because undetectable demagnetized magnets can be intermixed with actual magnets to allow rapid rotation of either type of magnets to be activated in one and the same device in a randomized protocol. Under a previously approved HMRI study protocol this new device has been shown to induce motor-evoked potentials (MEPs) in thenar muscles by highly focused stimulation of their cortical representation in the precentral gyrus.

In the present pilot study, the investigators would like to conduct a randomized double-blind placebo-controlled clinical trial to test the therapeutic effectiveness of bilateral mTMS stimulation of the supplementary motor areas (mTMS-SMA therapy) in TS patients presenting with tics uncontrolled by standard drug and behavioral treatment. The specifics aims of this study are:

1. To compare the immediate benefits obtained by TS patients subjected to two weeks of five day per week mTMS-SMA therapy with respect to those obtained by TS patients receiving placebo (sham stimulation) treatment, in terms of reduction of the frequency of tics and alleviation (primary end points) and of other comorbidities (ADHD and OCD, secondary end points) of TS.
2. To compare the long-term benefits as above over a two-month follow up period in the same set of treated and placebo control TS patients

The investigators will conduct this study in 20, English speaking, TS patients in the age range of 8 to 20 years. Half the patients will be randomly assigned in a double-blind manner to the active treatment or the placebo control (sham treatment) groups that will be appropriately age-and gender-matched. Randomization will be completed by the study team by alternating between cap A and cap B, within specific cohorts. The cohorts will be as follows: 8-13 years of age at time of enrollment and 14-20 years of age at time of enrollment. The stimulus parameters used will be those that are effective in upregulating the excitability of the motor pathways to elicit MEPs in the thenar muscles. The investigators believe that mTMS-SMA therapy will produce both short- and long-term benefit for TS patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 8 and 20 years old,
* A clinical diagnosis of TS as defined by the DSM V
* YGTSS score of 13 or more (performed at Visit 1).
* Patients with the following comorbidities: OCD, ADHD and anxiety disorders (as defined by the DSM V) will be allowed in the study. This will be assessed during Visit 1.
* The patients may be on medications for the treatment of TS or allowed comorbidities provided the medication regimen is stable for six weeks prior to inclusion in the study and remains unchanged for the 10 weeks that the study will last.

Exclusion Criteria:

* Any history of neurological, or psychiatric disorders including epilepsy and autism spectrum disorder, other than other than the allowed comorbidities (see above).
* An IQ less than 80, this will be assessed during Visit 1.
* Any changes in medications prescribed for the treatment of TS or allowed comorbidities six weeks prior to inclusion in the study or at any time during the study.
* The presence of metal implants or metallic devices in the head
* Any history of drug or alcohol abuse
* Any medication changes during the six weeks preceding enrollment or at any time during the 10-week course of the study

Ages: 8 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Change in tic severity from baseline to 2 months post-treatment | Day of first treatment session, End of weeks 1 and 2, as well as 1 month and 2 months after treatment
  The investigators will assess reduction in tics with the Yale Global Tic Severity Scale. It is a rating that is based on a clinician-rated, semistructured interview that begins with a systematic inquiry of tic symptoms in the preceding week. Five index scores are obtained: Total Motor Tic Score, Total Phonic Tic Score, Total Tic Score, Overall Impairment Rating, and Global Severity Score. The Total Motor Tic Score is derived by adding the five motor tics items (range = 0-25); the Total Phonic Tic Score is derived by adding the five phonic tics items (range = 0-25). The Total Tic Score is a summation of the Total Motor Tic and Total Phonic Tic Scores. The Overall Impairment Rating is rated on a 50-point scale anchored by 0 (No impairment) and 50 (Severe impairment). Finally, the Global Severity Score is a summation of the Total Motor Tic Score, Total Phonic Tic Score, and Overall Impairment Rating (range = 0-100). A higher score represents a worse outcome.

SECONDARY OUTCOMES:
Change in ADHD symptoms from baseline to two months post-treatment | Day of first treatment session, End of weeks 1 and 2, as well as 1 month and 2 months after treatment
  The investigators will assess if treatment had any effect on ADHD symptoms using the Vanderbilt ADHD Parent Rating Scale. This validated scale consists of 49 questions regarding frequency of behaviors and 2 about performance.
  Predominately inattentive subtype (6 of 9 behaviors), (scores of 2 or 3 are positive) on items 1-9, and a performance problem (scores of 1 or 2) in any item in the performance section.
  * Predominately hyperactive/Impulsive subtype requires 6 of 9 behaviors (scores of 2 or 3 are positive) on items 10-18 and a problem (1 or 2) in any item in the performance section.
  * The Combined Subtype requires the above criteria on both inattention and hyperactivity/impulsivity.
Change in OCD symptoms from baseline to two months post-treatment | Day of first treatment session, End of weeks 1 and 2, as well as 1 month and 2 months after treatment
  The investigators will assess if treatment had any effect on OCD symptoms using the Yale-Brown Obsessive Compulsive Scale (Y-BOCS). The Y-BOCS is a 10-item scale designed to measure the severity and type of symptoms in people with obsessive-compulsive disorder (OCD) over the past seven days. The symptoms assessed are obsessions and compulsions. This scale is useful in tracking OCD symptoms at intake and during/after treatment. Total Y-BOCS scores range from 0 to 40, with higher scores indicating greater severity of OCD symptoms. Scores on the obsession and compulsion subscales range from 0 to 20, but only the total Y-BOCS score is interpreted. Total scores can be split into five categories, based on severity of symptoms.
  Under 7 are likely to be subclinical, 8-15 are likely to have a mild case of OCD, 16-23 are likely to have a moderate case of OCD, 24-31 are likely to have a severe case of OCD, 32-40 are likely to have an extreme case of OCD.

CONTACTS AND LOCATIONS:
Overall Officials: Keith A Coffman, M.D., Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Robertson MM, Eapen V, Cavanna AE. The international prevalence, epidemiology, and clinical phenomenology of Tourette syndrome: a cross-cultural perspective. J Psychosom Res. 2009 Dec;67(6):475-83. doi: 10.1016/j.jpsychores.2009.07.010. PMID 19913651
- [Background] Termine C, Selvini C, Rossi G, Balottin U. Emerging treatment strategies in Tourette syndrome: what's in the pipeline? Int Rev Neurobiol. 2013;112:445-80. doi: 10.1016/B978-0-12-411546-0.00015-9. PMID 24295630
- [Background] Rossini PM, Rossi S. Transcranial magnetic stimulation: diagnostic, therapeutic, and research potential. Neurology. 2007 Feb 13;68(7):484-8. doi: 10.1212/01.wnl.0000250268.13789.b2. PMID 17296913
- See also: Transcranial Brain Stimulation With Rapidly Spinning High-Field Permanent Magnets — https://ieeexplore.ieee.org/document/7473846/